CLINICAL TRIAL: NCT00189137
Title: Phase II Evaluation of Ifosfamide Plus Doxorubicin & Filgrastim Versus Gemcitabine Plus Docetaxel & Filgrastim in the Treatment of Localized Poor Prognosis Soft Tissue Sarcoma
Brief Title: Evaluation of Side Effects and Relative Activity of Two Chemotherapy Regimens in the Treatment Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2004.010; HUM 44800 (Other: University of Michigan IRBMED)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Ifosfamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxorubicin and ifosfamide (Active Comparator)
  Interventions: Drug: ifosfamide and doxorubicin vs gemcitabine and docetaxel
- gemcitabine and docetaxel (Experimental)
  Interventions: Drug: ifosfamide and doxorubicin vs gemcitabine and docetaxel

INTERVENTIONS:
Drug: ifosfamide and doxorubicin vs gemcitabine and docetaxel — Arm 1 will consist of the two drug combination of doxorubicin and ifosfamide (with mesna) Treatment will be delivered over 3 days at 21 day intervals. Patients will receive filgrastim days 4-10 or peg-filgrastim on day 4 as a myeloid growth factor.
  Arm 2 will consist of the two drug combination of gemcitabine (day 1, 8) and docetaxel (day 8) repeated at 21 day intervals. Patients will receive filgrastim as a myeloid growth factor days 9-15 or peg-filgrastim on day 4.
  All patients will receive 4 cycles of chemotherapy unless there is unacceptable toxicity or disease progression that may adversely impact the surgical plan for complete resection.

SUMMARY:
The purpose of this study is to explore how a sarcoma is affected by and the side effects of a newer combination of chemotherapy drugs(gemcitabine and docetaxel)as compared to a standard combination of chemotherapy drugs, ifosfamide and doxorubicin.

DETAILED DESCRIPTION:
The purpose of this study is to explore the relative activity and toxicity of a newer combination of chemotherapy drugs, gemcitabine and docetaxel, as compared to a standard combination of chemotherapy drugs, ifosfamide and doxorubicin.

Ifosfamide and Doxorubicin, given in combination, are recognized as a standard of care for some types of sarcoma. Both gemcitabine and docetaxel are approved by the US Food and Drug Administration (FDA) for the treatment of some cancers (cancers of the pancreas, lung) because patients with those cancers treated with either gemcitabine or docetaxel experienced shrinkage of their tumor or improvement in their symptoms. However, neither gemcitabine or docetaxel is approved for sarcoma, but the combination of gemcitabine and docetaxel is a standard treatment for advanced sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* no evidence of metastasis
* soft tissue sarcoma
* intermediate or high histologic grade
* greater than 5 cm
* Zubrod performance status 1 or better
* age 10 or older

Exclusion Criteria:

* clear cell, alveolar soft part, Ewing's rhabdosarcoma, undifferentiated small cell or Kaposi's
* prior chemotherapy
* nephrectomy
* active unstable angina pectoris
* concurrent therapy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-08; Primary Completion 2012-11 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Schuetze, MD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Davis EJ, Zhao L, Lucas DR, Schuetze SM, Baker LH, Zalupski MM, Thomas D, Chugh R. SPARC expression in patients with high-risk localized soft tissue sarcoma treated on a randomized phase II trial of neo/adjuvant chemotherapy. BMC Cancer. 2016 Aug 20;16:663. doi: 10.1186/s12885-016-2694-2. PMID 27544129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 patients were enrolled and randomized at the University of Michigan, however 4 patients withdrew consent prior to treatment. 80 patients began study treatment.
Groups:
- Doxorubicin and Ifosfamide: Arm 1 will consist of the two drug combination of doxorubicin and ifosfamide (with mesna) Treatment will be delivered over 3 days at 21 day intervals. Patients will receive filgrastim days 4-10 or peg-filgrastim on day 4 as a myeloid growth factor.
  All patients will receive 4 cycles of chemotherapy unless there is unacceptable toxicity or disease progression that may adversely impact the surgical plan for complete resection.
- Gemcitabine and Docetaxel: Arm 2 will consist of the two drug combination of gemcitabine (day 1, 8) and docetaxel (day 8) repeated at 21 day intervals. Patients will receive filgrastim as a myeloid growth factor days 9-15 or peg-filgrastim on day 4.
  All patients will receive 4 cycles of chemotherapy unless there is unacceptable toxicity or disease progression that may adversely impact the surgical plan for complete resection.
Period: Overall Study
Arm/Group | Doxorubicin and Ifosfamide | Gemcitabine and Docetaxel
Started | 37 | 43
Completed | 37 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxorubicin and Ifosfamide | Gemcitabine and Docetaxel | Total
Number analyzed (Participants) | 37 | 43 | 80
Age, Continuous [Median (Full Range); unit: years] | 55 [19 to 76] | 57 [19 to 74] | 56 [19 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 22 | 31 | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Hospitalized in Each Arm.
Description: To contrast the proportion of treated patients hospitalized subsequent to treatment with gemcitabine and docetaxel as compared to doxorubicin and ifosfamide as neoadjuvant or adjuvant therapy of poor prognosis soft tissue sarcoma.
Time Frame: 12 weeks
Measure: Number; unit: percentage of patients hospitalized
Arm/Group | Doxorubicin and Ifosfamide | Gemcitabine and Docetaxel
Number analyzed (Participants) | 37 | 43
percentage of patients hospitalized | 35 | 26

2. Secondary Outcome: The Percentage of Patients Alive Without Disease at 2 Years
Description: Disease-free survival
Time Frame: 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Doxorubicin and Ifosfamide | Gemcitabine and Docetaxel
Number analyzed (Participants) | 37 | 43
percentage of patients | 57 | 74

ADVERSE EVENTS:
Arm/Group | Doxorubicin and Ifosfamide | Gemcitabine and Docetaxel
Serious Adverse Events (participants affected / at risk) | 12/37 | 12/43
Other Adverse Events (participants affected / at risk) | 30/37 | 33/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin and Ifosfamide (N=37) | Gemcitabine and Docetaxel (N=43)
Ataxia (incoordination) (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 1 | 0
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Edema: limb (General disorders) | 0 | 1
Fever (General disorders) | 0 | 2
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxorubicin and Ifosfamide (N=37) | Gemcitabine and Docetaxel (N=43)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 | 4
Ataxia (incoordination) (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 1 | 0
Cardiac troponin I (cTnI) (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 | 6
Hemoglobin (Blood and lymphatic system disorders) | 9 | 4
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 | 0
Infection with unknown ANC (Infections and infestations) | 1 | 0
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 25 | 7
Lymphopenia (Blood and lymphatic system disorders) | 8 | 5
Mucositis/stomatitis (clinical exam) (Investigations) | 1 | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 23 | 7
Pain (General disorders) | 1 | 2
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 4 | 0
Platelets (Blood and lymphatic system disorders) | 12 | 6
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 | 1
Syncope (fainting) (Nervous system disorders) | 1 | 1
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Edema: limb (General disorders) | 0 | 1
Fever (General disorders) | 0 | 2
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 0 | 1
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 0 | 1
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 | 5
Nausea (Gastrointestinal disorders) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes